CLINICAL TRIAL: NCT02453997
Title: Mycophenolic Acid Pharmacokinetics and Pharmacogenomics - Impact on the Clinical Outcomes of Patients With Severe Lupus Nephritis
Brief Title: Mycophenolic Acid Pharmacokinetics and Pharmacogenomics in Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: United Christian Hospital (Other)
Responsible Party: Principal Investigator, Dr. Desmond Yat-Hin Yap, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW12-462
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; mycophenolic acid; pharmacokinetics; pharmacogenomics
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples for pharmacogenomics analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study investigate mycophenic acid (MPA) pharmacokinetics and pharmacogenomics and their impact on the clinical outcomes in lupus nephritis (LN) patients. Lupus nephritis patients (both active or inactive) will be recruited. MPA levels will be checked at 1, 2, 4, 8, 10, 12 hrs after MMF administration by an enzymatic assay upon recruitment, then at 6-months' intervals and also when clinically significant events occurred. The MPA levels will be correlated with clinical parameters and outcomes. Pharmacogenomics studies will also be carried out and correlated with MPA exposure and clinical outcomes.

DETAILED DESCRIPTION:
This study investigate mycophenic acid (MPA) pharmacokinetics and pharmacogenomics and their impact on the clinical outcomes in lupus nephritis (LN) patients. Lupus nephritis patients (both active or inactive) will be recruited. MPA levels will be checked at 1, 2, 4, 8, 10, 12 hrs after MMF administration by an enzymatic assay upon recruitment, then at 6-months' intervals and also when clinically significant events occurred. The MPA levels will be correlated with clinical parameters and outcomes. For active patients, the MPA levels will be correlated with treatment response (CR or PR) and side effects. For patients in remission, the MPA levels will be correlated with drug tolerability and relapse. Pharmacogenomics studies will also be carried out and correlated with MPA exposure and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recent active LN (biopsy-proven Class III/IV+/-V LN according to the ISN/RPS 2003 classifications within 3 months, with proteinuria >0.5 g/day and/or active urinary sediments) who receive corticosteroids and MMF (1g bd for 6 months) as induction treatment.
2. LN patients in remission (defined as proteinuria <0.5 g/day with inactive urinary sediment, prednisolone <10 mg/day) and on stable MMF maintenance (dose unchanged within the previous 3 months).

Exclusion Criteria:

1. Patients who receive enteric-coated mycophenolic acid (myfortic).
2. Patients who receive concomitant calcineurin inhibitors (e.g. cyclosporine or tacrolimus) other than corticosteroids and MMF.
3. Patients who receive concomitant medications which affect the MPA pharmacokinetics such as cholestyramine, acyclovir, and rifampicin.
4. Patients who are pregnant or lactating.
5. Patients with gastric emptying disorders
6. Patients with hepatic or biliary diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lupus Nephritis patients (both active or remission)
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
AUC (0-12) | 24 months

SECONDARY OUTCOMES:
Infection | 24 months
Gastrointestinal disturbances | 24 months
Complete or partial remission | 24 months
Relapse | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - United Christian Hospital, Hong Kong